CLINICAL TRIAL: NCT03209206
Title: The Effectiveness and Safety of Intravesical Docetaxel Instillation After Operation to Prevent Intravesical Recurrence After Radical Nephroureterectomy or Distal Ureterectomy in Upper Urinary Tract Urothelial Carcinoma: A Prospective Study
Brief Title: The Effectiveness and Safety of Intravesical Docetaxel Instillation for Prevent Bladder Recurrence
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ja Hyeon Ku, Professor, MD., PHD., Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SeoulNUHUro
Record Dates: First submitted 2017-06-30; First posted 2017-07-06 (Actual); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Urothelial Carcinoma
Keywords: Intravesical Chemotherapy; Docetaxel; Radical Nephroureterectomy
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — Docetaxel

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Phase II Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Docetaxel bladder instillation arm (Experimental): After Surgery, intravesical chemotherapy with in 48 hrs (Docetaxel 75 mg diluted in 100 cc of normal saline)
  Interventions: Drug: Docetaxel
- Control arm (Placebo Comparator): After Surgery, intravesical chemotherapy with in 48 hrs (Placebo, 100 cc of normal saline)
  Interventions: Drug: Placebo Normal saline

INTERVENTIONS:
Drug: Docetaxel — Intravesical Instillation of Docetaxel (Docetaxel 75 mg diluted in 100 cc of normal saline) after operation of Upper urinary tract urothelial carcinoma (With in 48 hrs)
  Other Names: Instillation docetaxel after radical nephroureterectomy
  Arms: Docetaxel bladder instillation arm
Drug: Placebo Normal saline — Intravesical Instillation of Normal saline (100 cc of normal saline) after operation of Upper urinary tract urothelial carcinoma (With in 48 hrs)
  Other Names: Instillation Normal saline after radical nephroureterectomy
  Arms: Control arm

SUMMARY:
The investigators evaluated the efficacy of a single early intravesical instillation of doxetaxel in the prevention of bladder recurrence after nephroureterectomy or distal ureterectomy for upper urinary tract urothelial carcinoma (UUT-UC).

DETAILED DESCRIPTION:
Approximately 20% to 50% of patients with upper urinary tract urothelial carcinoma (UUT-UC) experience bladder recurrence after nephroureterectomy. Although many agents have been administered for the prevention of bladder recurrence, the standard prophylactic treatment has yet to be established. A meta-analysis found that a single instillation of chemotherapy immediately after transurethral resection of bladder tumor (TURBT) significantly decreased the risk of recurrence in patients with bladder cancer. Indeed, a single early instillation of Docetaxel was found to reduce the post-TURBT bladder recurrence rate among patients with bladder cancer.

In this prospective, randomized study, the investigators evaluated the efficacy of a single, early, intravesical instillation of Docetaxel in the prevention of bladder recurrence after nephroureterectomy for UUT-UC.

ELIGIBILITY:
Inclusion Criteria:

* Upper urinary tract urothelial cell carcinoma
* Hb>10g/dL, ANC >1500mm3, Platelet > 100K
* Total bilirubin : 1.5 times lower than the normal upper limit
* AST/ALT: 1.8 times lower than the normal upper limit
* Alkaline phosphatase: 1.8 times lower than the normal upper limit

Exclusion Criteria:

* Concomitant bladder tumor
* Patients diagnosed with bladder cancer within the last 3 years
* Previous history of hypersensitivity to Docetaxel
* Neurogenic Bladder
* Patients who received chemotherapy for cancer within the last 6 months
* Patients with active disease not fit for this study
* ANC <1500mm3
* Pregnant or lactating women
* Patients with severe hepatic dysfunction
* patients with severe renal impairment
* patients with hypersensitivity to mannitol, paraplatin, platinum compounds
* Patients with complications of infection
* Patients suspected of having infectious fever

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2017-06-28 (Actual); Primary Completion 2020-06-19 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence in bladder | 2years
  Present of bladder recurrence after intervention in follow up cystoscopy or CT scan

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 2years
  Present of adverse event after intervention
Overall Survival | 2years
  Overall Survival rate during follow up period
Time to recurrence | 2years
  Time to bladder recurrence after intervention in follow up cystoscopy or CT scan

CONTACTS AND LOCATIONS:
Overall Officials: Ja Hyeon Ku, M.D.,PH.D, Study Director — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ito A, Shintaku I, Satoh M, Ioritani N, Aizawa M, Tochigi T, Kawamura S, Aoki H, Numata I, Takeda A, Namiki S, Namima T, Ikeda Y, Kambe K, Kyan A, Ueno S, Orikasa K, Katoh S, Adachi H, Tokuyama S, Ishidoya S, Yamaguchi T, Arai Y. Prospective randomized phase II trial of a single early intravesical instillation of pirarubicin (THP) in the prevention of bladder recurrence after nephroureterectomy for upper urinary tract urothelial carcinoma: the THP Monotherapy Study Group Trial. J Clin Oncol. 2013 Apr 10;31(11):1422-7. doi: 10.1200/JCO.2012.45.2128. Epub 2013 Mar 4. PMID 23460707
- [Result] Delto JC, Kobayashi T, Benson M, McKiernan J, Abate-Shen C. Preclinical analyses of intravesical chemotherapy for prevention of bladder cancer progression. Oncotarget. 2013 Feb;4(2):269-76. doi: 10.18632/oncotarget.852. PMID 23563166
- [Result] Wu P, Zhu G, Wei D, Liu S, Walsh K, Li D, Harron U, Wang X, Ma H, Wan B, Sun L, Yang Z, Wang J. Prophylactic intravesical chemotherapy decreases bladder tumor recurrence after nephroureterectomy for primary upper tract urothelial carcinoma: A systematic review and meta-analysis. J BUON. 2015 Sep-Oct;20(5):1229-38. PMID 26537069
- [Result] Laudano MA, Barlow LJ, Murphy AM, Petrylak DP, Desai M, Benson MC, McKiernan JM. Long-term clinical outcomes of a phase I trial of intravesical docetaxel in the management of non-muscle-invasive bladder cancer refractory to standard intravesical therapy. Urology. 2010 Jan;75(1):134-7. doi: 10.1016/j.urology.2009.06.112. Epub 2009 Nov 13. PMID 19913890
- [Result] Lu S, Neoh KG, Kang ET, Mahendran R, Chiong E. Mucoadhesive polyacrylamide nanogel as a potential hydrophobic drug carrier for intravesical bladder cancer therapy. Eur J Pharm Sci. 2015 May 25;72:57-68. doi: 10.1016/j.ejps.2015.03.006. Epub 2015 Mar 13. PMID 25772330
- [Result] Barlow L, McKiernan J, Sawczuk I, Benson M. A single-institution experience with induction and maintenance intravesical docetaxel in the management of non-muscle-invasive bladder cancer refractory to bacille Calmette-Guerin therapy. BJU Int. 2009 Oct;104(8):1098-102. doi: 10.1111/j.1464-410X.2009.08543.x. Epub 2009 Apr 15. PMID 19389012